CLINICAL TRIAL: NCT03526874
Title: Occipital Nerve Blocks for Acute Treatment of Pediatric Migraine
Brief Title: Occipital Blocks for Acute Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-014939; K23NS102521 (NIH)
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Migraine, Headache; Episodic Migraine
Keywords: Pain; Chronic Migraine; Episodic Migraine; Headache; Nerve Block
MeSH Terms: conditions — Headache; Pain | interventions — Lidocaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind greater occipital nerve injection of lidocaine versus saline after open-label lidocaine cream run-in
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Greater Occipital Nerve (GON) Block with Lidocaine (Experimental): Subjects randomized to this arm receive 2 mL injection of lidocaine 2% over the right and left greater occipital nerve at the baseline study visit.
  All subjects then complete daily headache-related questions through a Headache Diary and other assessments for 28 days.
  Interventions: Drug: Lidocaine 4% Topical Application Cream [LMX 4]; Drug: Lidocaine Hydrochloride 2 mg/mL Injectable Solution
- Greater Occipital Nerve (GON) Block with Saline (Placebo Comparator): Subjects randomized to this arm receive 2 mL injection of preservative-free normal saline over the right and left greater occipital nerve at the baseline study visit.
  All subjects then complete daily headache-related questions through a Headache Diary and other assessments for 28 days.
  Interventions: Drug: Lidocaine 4% Topical Application Cream [LMX 4]; Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine 4% Topical Application Cream [LMX 4] — Run-in Step: All subjects receive 32 mg (4 cm ribbon of cream) applied, bilaterally, over greater occipital nerve.
Drug: Lidocaine Hydrochloride 2 mg/mL Injectable Solution — Subjects, who continue to experience headache pain after the run-in step, receive 2 (2 mL) injections of the active treatment.
  Arms: Greater Occipital Nerve (GON) Block with Lidocaine
Drug: Normal Saline — Subjects, who continue to experience headache pain after the run-in step, receive 2 (2 mL) injections of the comparator.
  Other Names: 0.9% Sodium Chloride
  Arms: Greater Occipital Nerve (GON) Block with Saline

SUMMARY:
Migraine affects 10-28% of children and adolescents and yet 20-30% of patients are ineffectively treated with current oral and nasal options. Peripheral nerve blocks (PNBs), injections of local anesthetics over branches of the occipital and/or trigeminal nerves, have been associated with possible benefit for pediatric headaches in case series, and may be useful for both acute and preventive treatment of migraine for children who fail less invasive treatments. In fact, 80% of pediatric headache specialists reported using peripheral nerve blocks and carry low risk of serious side effects; however, peripheral nerve blocks have never been tested, formally, in a randomized pediatric trial.

By applying a novel design that utilizes lidocaine cream as a run-in step, investigators intend to test the efficacy of the most commonly used peripheral nerve block, the greater occipital nerve (GON) block, as an acute treatment for pediatric migraine and determine whether lidocaine cream leads to successful blinding of the injection.

The GON block is expected to prove effective in decreasing the pain of migraine, with lidocaine being superior to saline and lidocaine cream maintaining blinding.

DETAILED DESCRIPTION:
There are two substantial hurdles that must be overcome in designing a trial to test the efficacy of PNBs: high placebo response rate and possible unblinding. In order to test the efficacy of this commonly used treatment for children and adolescents with difficult-to-treat headache, we need utilize a trial design which will address the high placebo response rate and the potential lack of blinding.

About 194 children, recruited over a 3.5 year period at Children's Hospital of Philadelphia, will take part in this study. Participation will last about one month and involve one in-person study visit, and then completion of headache-related surveys, at home, for 28 days. Lidocaine cream lead-in will be used open-label for all subjects followed by double-blind randomized injections of active treatment (lidocaine) versus comparator (saline) in subjects who continue to have significant headache.

To accomplish our secondary objectives, we will examine how expectation is affected by perceived treatment, and how expectations, measured in patients, parents, and providers, influence outcomes in pediatric and adolescent acute migraine.

ELIGIBILITY:
Inclusion Criteria:

* Children / Adolescents:

  * Males or females, ages 7 - 21, of any gender, race, or ethnicity
  * Diagnosis of episodic or chronic migraine with acute headache flare lasting up to 3 months unresponsive to acute medications. Patients who report that acute medications were not used during this headache flare because those medications have been ineffective for several prior headache flares will be included
  * Informed parental consent and subject assent
  * Girls, who have reached menarche, must have a negative urine or serum pregnancy test
  * Weight > 25kg
* Parents:

  * Parents or guardians of children enrolled, who speak either English or Spanish, and provide parental/guardian permission (informed consent) for their own participation
  * Subject (child) assent

Exclusion Criteria:

* Children / Adolescents:

  * Previous nerve block less than 3 months ago or more than 2 previous nerve blocks
  * Allergy to local anesthetics
  * Skull defect or break in the skin at the planned site of cream application or GON injection
  * Any investigational drug use within 30 days prior to enrollment, or 90 days prior to enrollment for medications targeted at Calcitonin Gene-Related Peptide
  * Pregnant or lactating females
  * Parents/guardians or subjects who, in the opinion of the Investigator, may be non- compliant with study schedules or procedures
  * Significant adverse event with prior injection or procedure
  * New abnormalities on physical or neurological examination
  * Newly reported red flags in headache history which prompt investigation for secondary headache
  * Non-English and Non-Spanish speaking
  * Non-English speaking with no Spanish interpreter available
* Parents:

  * Parents or guardians of children enrolled, who do not speak either English or Spanish
  * Parental/guardian permission and/or subject (child) assent has been declined
  * Parents or guardians, who in the opinion of the investigator, may be non-compliant or unable to complete the questionnaires

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L. Szperka, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia and Perelman School of Medicine at the University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hershey AD, Powers SW, Vockell AL, LeCates S, Kabbouche MA, Maynard MK. PedMIDAS: development of a questionnaire to assess disability of migraines in children. Neurology. 2001 Dec 11;57(11):2034-9. doi: 10.1212/wnl.57.11.2034. PMID 11739822
- [Background] Powers SW, Patton SR, Hommel KA, Hershey AD. Quality of life in childhood migraines: clinical impact and comparison to other chronic illnesses. Pediatrics. 2003 Jul;112(1 Pt 1):e1-5. doi: 10.1542/peds.112.1.e1. PMID 12837897
- [Background] Split W, Neuman W. Epidemiology of migraine among students from randomly selected secondary schools in Lodz. Headache. 1999 Jul-Aug;39(7):494-501. doi: 10.1046/j.1526-4610.1999.3907494.x. PMID 11279934
- [Background] Abu-Arefeh I, Russell G. Prevalence of headache and migraine in schoolchildren. BMJ. 1994 Sep 24;309(6957):765-9. doi: 10.1136/bmj.309.6957.765. PMID 7950559
- [Background] Szperka CL, Gelfand AA, Hershey AD. Patterns of Use of Peripheral Nerve Blocks and Trigger Point Injections for Pediatric Headache: Results of a Survey of the American Headache Society Pediatric and Adolescent Section. Headache. 2016 Nov;56(10):1597-1607. doi: 10.1111/head.12939. Epub 2016 Oct 12. PMID 27731894
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were contacted over the phone and, if interested, verbally consented and prescreened. Potentially eligible subjects were schedule for a visit. After signing consent during the study visit, eligibility was assessed. Approximately 438 patients were prescreened, and we have approached 140. Of those 63 were recruited and 58 randomized (5 screen failed after consent)).
Pre-assignment Details: Lidocaine cream lead in. If the subject responded to lidocaine cream application after 30 minutes they were not randomized. All eligible subjects were randomized.
Groups:
- Greater Occipital Nerve (GON) Block With Lidocaine: Subjects randomized to this arm receive 2 mL injection of lidocaine 2% over the right and left greater occipital nerve at the baseline study visit.
  All subjects then complete daily headache-related questions through a Headache Diary and other assessments for 28 days.
  Lidocaine 4% Topical Application Cream [LMX 4]: Run-in Step: All subjects receive 32 mg (4 cm ribbon of cream) applied, bilaterally, over greater occipital nerve.
  Lidocaine Hydrochloride 2 mg/mL Injectable Solution: Subjects, who continue to experience headache pain after the run-in step, receive 2 (2 mL) injections of the active treatment.
- Greater Occipital Nerve (GON) Block With Saline: Subjects randomized to this arm receive 2 mL injection of preservative-free normal saline over the right and left greater occipital nerve at the baseline study visit.
  All subjects then complete daily headache-related questions through a Headache Diary and other assessments for 28 days.
  Lidocaine 4% Topical Application Cream [LMX 4]: Run-in Step: All subjects receive 32 mg (4 cm ribbon of cream) applied, bilaterally, over greater occipital nerve.
  Normal Saline: Subjects, who continue to experience headache pain after the run-in step, receive 2 (2 mL) injections of the comparator.
Period: Overall Study
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.80 (2.00) | 16.19 (1.52) | 16.00 (1.80)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants' self-representation of gender identity
  Participants
    Gender: Female | 21 | 23 | 44
    Gender: Male | 8 | 3 | 11
    Gender: Non-binary | 0 | 2 | 2
    Gender: Other | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Participants' classification as male or female based on biological distinctions
  Participants
    Female | 21 | 26 | 47
    Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 24 | 24 | 48
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
Migraine Diagnosis [Count of Participants; unit: Participants]
  Episodic Migraine | 13 | 14 | 27
  Chronic migraine | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Numeric Analog Scale (NRS)
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Numeric Rating Scale (NRS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. NRS scale is a 0 to 10 scale, with 0 meaning no pain and 10 meaning "the worse pain imaginable". A mean change of 2-points has been shown to be clinically relevant.
Time Frame: Pre-injection (*Baseline*) and 30 minutes Post-injection
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
score on a scale | 2.3 (1.9) | 1.1 (1.9)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.013, t-test, 2 sided

2. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Visual Analog Scale (VAS)
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Visual Analog Scale (VAS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. VAS scale is a 0 to 100 visual scale, with 0 meaning no pain and 100 meaning "the worse pain imaginable".
Time Frame: Pre-injection and 30 minutes Post-injection
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
score on a scale | 24.97 (4.09) | 12.86 (3.61)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.031, t-test, 2 sided

3. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Numeric Analog Scale (NRS) by Sex
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Numeric Rating Scale (NRS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. By sex. NRS scale is a 0 to 10 scale, with 0 meaning no pain and 10 meaning "the worse pain imaginable". A mean change of 2-points has been shown to be clinically relevant.
Time Frame: Pre-injection (*Baseline*) and 30 minutes Post-injection
Population: Overall number is divided between the different sex subcategories for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
score on a scale
  Female: number analyzed (Participants) | 21 | 26
  Female | 2.5 (2) | 1 (1.8)
  Male: number analyzed (Participants) | 8 | 3
  Male | 2 (1.8) | 2 (2)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.0162, ANOVA; Two-way Anova to test sex interaction with treatment effect. The study was not powered for subgroup analyses

4. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Visual Analog Scale (VAS) by Sex
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Visual Analog Scale (VAS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. By sex. VAS scale is a 0 to 100 visual scale, with 0 meaning no pain and 100 meaning "the worse pain imaginable".
Time Frame: Pre-injection and 30 minutes Post-injection
Population: Overall number is divided between the different sex subcategories for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
score on a scale
  Female: number analyzed (Participants) | 21 | 26
  Female | 25.5 (23) | 12 (19.6)
  Male: number analyzed (Participants) | 8 | 3
  Male | 23.6 (20.6) | 10.3 (19)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.04, ANOVA — Two-way Anova to test sex interaction with treatment effect. The study was not powered for subgroup analyses

5. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Numeric Analog Scale (NRS) by Ethnicity
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Numeric Rating Scale (NRS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. By ethnicity. NRS scale is a 0 to 10 scale, with 0 meaning no pain and 10 meaning "the worse pain imaginable". A mean change of 2-points has been shown to be clinically relevant.
Time Frame: Pre-injection (*Baseline*) and 30 minutes Post-injection
Population: Overall number is divided between the different ethnic subcategories for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 28
score on a scale
  Hispanic: number analyzed (Participants) | 4 | 2
  Hispanic | 1.3 (1.5) | -0.5 (0.7)
  Non-Hispanic: number analyzed (Participants) | 25 | 26
  Non-Hispanic | 2.5 (2) | 1.2 (1.9)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.0098, ANOVA; Two-way Anova to test ethnicity interaction with treatment effect. The study was not powered for subgroup analyses

6. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Visual Analog Scale (VAS) by Ethnicity
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Visual Analog Scale (VAS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. By ethnicity. VAS scale is a 0 to 100 visual scale, with 0 meaning no pain and 100 meaning "the worse pain imaginable".
Time Frame: Pre-injection and 30 minutes Post-injection
Population: Overall number is divided between the different ethnic subcategories for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 28
score on a scale
  Hispanic: number analyzed (Participants) | 4 | 2
  Hispanic | 9 (14.4) | -3.5 (4.9)
  Non-Hispanic: number analyzed (Participants) | 25 | 26
  Non-Hispanic | 27.5 (22.2) | 14.5 (19.8)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.02, ANOVA; Two-way Anova to test ethnicity interaction with treatment effect. The study was not powered for subgroup analyses

7. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Numeric Analog Scale (NRS) by Race
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Numeric Rating Scale (NRS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. By race. NRS scale is a 0 to 10 scale, with 0 meaning no pain and 10 meaning "the worse pain imaginable". A mean change of 2-points has been shown to be clinically relevant.
Time Frame: Pre-injection (*Baseline*) and 30 minutes Post-injection
Population: Overall number is divided between the different race subcategories for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
score on a scale
  Asian: number analyzed (Participants) | 1 | 1
  Asian | 0 (0) | 0 (0)
  Black: number analyzed (Participants) | 2 | 3
  Black | 4 (2.8) | 2 (2.6)
  White: number analyzed (Participants) | 24 | 24
  White | 2.4 (1.9) | 0.8 (1.6)
  Multiple races: number analyzed (Participants) | 2 | 1
  Multiple races | 1 (1.4) | 5 (0)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.01, ANOVA; Two-way Anova to test race interaction with treatment effect. The study was not powered for subgroup analyses

8. Primary Outcome: Mean Change in Pain Intensity Scores Measured by the Visual Analog Scale (VAS) by Race
Description: By subtracting the 30 minutes post-injection score from the pre-injection score, measured on a Visual Analog Scale (VAS), the mean change, in the lidocaine versus saline groups, will be used as the primary outcome measure. By race. VAS scale is a 0 to 100 visual scale, with 0 meaning no pain and 100 meaning "the worse pain imaginable".
Time Frame: score on a scale
Population: Overall number is divided between the different race subcategories for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
score on a scale
  Asian: number analyzed (Participants) | 1 | 1
  Asian | -12 (0) | 3 (0)
  Black: number analyzed (Participants) | 2 | 3
  Black | 26 (26.9) | 21.3 (11.7)
  White: number analyzed (Participants) | 24 | 24
  White | 27.2 (21.6) | 10 (17.4)
  Multiple races: number analyzed (Participants) | 2 | 1
  Multiple races | 14 (21.2) | 66 (0)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.0329, ANOVA; Two-way Anova to test race interaction with treatment effect. The study was not powered for subgroup analyses

9. Secondary Outcome: Change From Baseline Disability
Description: The PedMIDAS will assess changes in functional disability due to headache. The PedMIDAS is a validated 6-question scale that captures headache-related disability-across multiple domains of functioning including school, home, social, and recreational-for pediatric and adolescent aged patients over 3 months. The instrument measures the number of days in which subjects missed activities due to headache or migraine. The measure yields a total score by summing items ranging from 0 to 90 day. The higher the score the higher the disability. Change in total score (total at week 4 minus total at baseline) is reported.
Time Frame: Baseline and Week 4
Population: Missing values were omitted from testing.
Measure: Mean (Standard Error); unit: change of score on a scale
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 28 | 25
change of score on a scale | 0.036 (8.46) | -13.36 (9.39)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.294, t-test, 2 sided

10. Secondary Outcome: Change From Baseline Disability to Day 7
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (Short Form) will assess changes in functional disability due to headache. The PROMIS Pain Interference (Short Form) measures the self-reported consequences of pain on relevant aspects of the subject's life over the past seven days. A pain item pool was developed to yield scores on a T-score scale with a mean of 50 and standard deviation of 10. A higher PROMIS T-score represents more pain interference, a T-score of 60 is one standard deviation (SD) worse than average. By comparison, a pain interference T-score of 40 is one SD better than average.
Time Frame: Baseline and Day 7
Population: Missing values were omitted from testing.
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 28 | 24
t-score | 5.78 (1.54) | 2.11 (1.09)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.058, t-test, 2 sided

11. Secondary Outcome: Change From Baseline Disability to Week 4
Description: The PROMIS Pain Interference (Short Form) will assess changes in functional disability due to headache. The PROMIS Pain Interference (Short Form) measures the self-reported consequences of pain on relevant aspects of the subject's life over the past seven days. A pain item pool was developed to yield scores on a T-score scale with a mean of 50 and standard deviation of 10. A higher PROMIS T-score represents more pain interference, a T-score of 60 is one SD worse than average. By comparison, a pain interference T-score of 40 is one SD better than average.
Time Frame: Baseline and Week 4
Population: Missing values were omitted from testing.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 28 | 25
T-score | 5.05 (1.75) | 2.06 (1.35)
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.182, t-test, 2 sided

12. Secondary Outcome: Percentage of Subjects With Pain Freedom
Description: The measurement involves resolution of headache pain within 30 minutes after injection and prior to any rescue medications. Data will be collected prospectively from subjects, at the study visit.
Time Frame: 30 minutes Post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
Participants | 5 | 2
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.423, Fisher Exact

13. Secondary Outcome: Percentage of Subjects With Pain Relief or Headache Response
Description: The measurement involves improvement in headache from "severe or moderate" to "none or mild" within 30 minutes and before any rescue medications. Data will be collected prospectively from subjects at the study visit.
Time Frame: 30 minutes Post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
Participants | 15 | 7
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.030, Chi-squared

14. Secondary Outcome: Percentage of Subjects With Sustained Pain Freedom
Description: The measurement involves being pain-free within 30 minutes and lasting at least 24 hours, with no use of rescue medication and no relapse or recurrence. Data will be collected prospectively from subjects, via text, in an electronic headache diary.
Time Frame: 24 hours Post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
Participants | 4 | 0
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.112, Fisher Exact

15. Secondary Outcome: Percentage of Subjects With Sustained Pain Relief
Description: The measurement involves having pain-relief within 30 minutes and lasting at least 24 hours, with no use of rescue medication and no relapse or recurrence. Data will be collected prospectively from subjects, via text, in an electronic headache diary.
Time Frame: 24 hours Post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
Participants | 7 | 1
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.052, Fisher Exact

16. Secondary Outcome: Percentage of Subjects With Freedom From All Symptoms of Migraine
Description: The presence or absence of photophobia, phonophobia, and nausea will be collected from subjects prospectively, via text, in an electronic headache diary.
Time Frame: 24 hours Post-injection
Measure: Count of Participants; unit: Participants
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
Number analyzed (Participants) | 29 | 29
Participants | 14 | 6
Statistical Analysis 1: Comparison: Greater Occipital Nerve (GON) Block With Lidocaine vs Greater Occipital Nerve (GON) Block With Saline; Test type: Superiority; p = 0.027, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of the lead in treatment (lidocaine cream) application until 28days post-visit, *up to 29 days*.
Description: AEs were collected by RedCap survey, contact with the family and Epic chart review up until 28 days post visit. Serious adverse events (SAEs) were reported to the Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) within 24h of knowledge of the event. AEs were reported to the IRB at the next continuing review.
Arm/Group | Greater Occipital Nerve (GON) Block With Lidocaine | Greater Occipital Nerve (GON) Block With Saline
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/29
Other Adverse Events (participants affected / at risk) | 29/29 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Greater Occipital Nerve (GON) Block With Lidocaine (N=29) | Greater Occipital Nerve (GON) Block With Saline (N=29)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) — Participant reported insufficient relief after study nerve block. After nerve block with open-label lidocaine she developed symptoms of anaphylaxis, and was treated with epinephrine and albuterol. She was observed in the ED and symptoms resolved.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Greater Occipital Nerve (GON) Block With Lidocaine (N=29) | Greater Occipital Nerve (GON) Block With Saline (N=29)
Pre-syncope/syncope (General disorders) | 2 | 3
Confusion (Nervous system disorders) | 0 | 1
Worse headache pain (Nervous system disorders) | 21 | 26
Feeling dizzy (Nervous system disorders) | 21 | 21
Feeling sick to your stomach (Gastrointestinal disorders) | 16 | 20
Feeling worried or panicky (Nervous system disorders) | 17 | 21
Numbness (Nervous system disorders) | 18 | 11
Rash (Immune system disorders) | 1 | 1
Injection site problems (Injury, poisoning and procedural complications) | 8 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/74/NCT03526874/Prot_SAP_003.pdf
  • Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03526874/ICF_002.pdf